CLINICAL TRIAL: NCT00237484
Title: Effect of Infliximab in Hepatitis-C Genotype 1 Naïve Patients With High TNF-alpha on the Efficacy of Pegylated Interferon Alfa-2b/Ribavirin Therapy
Brief Title: Effect of Infliximab on the Efficacy of Peg-Intron/Ribavirin in Patients With Hepatitis C (Study P04257AM4)(COMPLETED)
Acronym: Pegade
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04257
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C, Chronic
Keywords: pegylated interferon alfa-2b; ribavirin; infliximab; chronic hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Remicade induction dose at Day -7 prior to initiation of PEGETRON treatment for up to 48 weeks
  Interventions: Drug: Induction dose of (a) infliximab followed by combination of (b) pegylated interferon alfa-2b and (c) ribavirin
- Arm B (Active Comparator): PEGETRON treatment for up to 48 weeks
  Interventions: Drug: Combination of (a) pegylated interferon alfa-2b and (b) ribavirin

INTERVENTIONS:
Drug: Induction dose of (a) infliximab followed by combination of (b) pegylated interferon alfa-2b and (c) ribavirin — 1. Powder for intravenous infusion (100 mg strength), intravenous, single dose of 5 mg/kg, at Day -7, prior to initiation of the following combination therapy:
  2. powder for injection in vials or Redipen (80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  3. 200 mg capsules, oral, dose of 800-1400 mg (weight based dosing as per PEGETRON Product Monograph), daily for up to 48 weeks
  Other Names: (a) SCH 215596, Remicade; PEGETRON combination therapy; (b) SCH 54031, PEG-Intron, PegIntron; (c) SCH 18908, REBETOL
  Arms: Arm A
Drug: Combination of (a) pegylated interferon alfa-2b and (b) ribavirin — 1. Powder for injection in vials or Redipen (80, 100, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  2. 200 mg capsules, oral, dose of 800-1400 mg (weight based dosing as per PEGETRON Product Monograph), daily for up to 48 weeks
  Other Names: PEGETRON combination therapy; (a) SCH 54031, PEG-Intron; PegIntron; (b) SCH 18908, REBETOL
  Arms: Arm B

SUMMARY:
This is a Phase IIIB, randomized, prospective, multicenter, single-country, open-label, controlled pilot trial designed to evaluate the effect of infliximab induction therapy on sustained virologic response (SVR) to treatment with pegylated interferon alfa-2b plus ribavirin in a group of 96 therapy-naïve subjects with genotype 1 hepatitis C virus (HCV) infection and high serum tumor necrosis factor (TNF)-alpha values.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be 18 to 65 years of age.
* HCV genotype 1 (including mixtures of subtypes of genotype 1).
* Naïve to interferon (any formulation) and ribavirin.
* Serum TNF-alpha >300 pg/mL(single measure at Pre-Screen Visit).
* HCV ribonucleic acid (RNA) positive.
* Any alanine aminotransferase (ALT) level.
* Fasting glucose should be 3.8-6.2 mmol/L. Results between 6.3-7.8 mmol/L require a HbA1c <=8.5%. All diabetic subjects must have an HbA1c <=8.5%, whether on medication or diet controlled.
* Liver biopsy within 24 months of enrolment demonstrating Stage 0-3 fibrosis (Metavir System).
* Compensated liver disease with the following minimum hematological, biochemical, and serological criteria at the screen visit (WNL = within normal limits):

  * Hemoglobin values of equal or more than 12 g/dL for females and 13 g/dL for males.
  * White blood cell (WBC) count equal to or more than 3,000/mm**3
  * Neutrophil count equal to or more than 1,500/mm**3
  * Platelet count equal to or more than 80,000/mm**3
  * Total bilirubin WNL
  * Indirect bilirubin WNL (unless non-hepatitis related factors such as Gilbert's disease explain an indirect bilirubin rise). In such cases indirect bilirubin should be less than or equal to 50 µmol/L
  * Albumin WNL
  * Serum creatinine WNL
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be willing to use an acceptable method of birth control, deemed acceptable by the investigator, (e.g., hormonal contraceptive, medically prescribed intrauterine device (IUD), condom in combination with spermicidal) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must understand and be able to adhere to the dosing and visit schedules, and agree to record, study medication compliance, concomitant medications, and adverse events accurately and consistently in a daily diary.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects who have used any investigational product within 30 days prior to enrollment.
* Acute HCV infection defined as infection for <6 months.
* Male partners to/or Heterosexually active women of childbearing potential not practicing a highly effective form of contraception.
* Positive screening for tuberculosis (TB) or Tuberculin Skin Test > 5mm.
* History or presence of cirrhosis (Stage 4 on Metavir System) and/or complication such as ascites, bleeding varices or hepatic encephalopathy
* Active hepatitis B virus (HBV) infection (hepatitis B surface antigen [HBsAg] positive).
* Any known pre-existing psychiatric condition that could interfere with the subject's participation in and completion of the study such as:

  * Pre-existing psychiatric condition, including but not limited to moderate to severe depression, or a history of severe psychiatric disorders, such as psychosis, suicidal ideation and/or suicidal attempt
  * Severe depression includes the following:

    * Hospitalization for depression,
    * Electro convulsive therapy for depression, or
    * Depression that resulted in a prolonged absence from work and/or significant disruption of daily functions.
* Subjects with uncontrolled hypertension and/or diabetes.
* Alcohol consumption >50 g/day.
* Nonprescription injection drug use in past 6 months.
* HIV antibody positive.
* Previous Infliximab or other anti-TNF treatment, previous interferon; Pegylated interferon alfa-2b and ribavirin of any form.
* Clinically significant impairment in cardiac or renal function, central nervous system, pulmonary, immunological, vascular and gastrointestinal disease.
* Current malignancy (other than resected cutaneous basal, squamous cell carcinoma and/or in situ cervical cancer).
* Use of illicit drugs which, in the investigator's opinion, may interfere with compliance with the study procedures.
* Any other condition which, in the opinion of a physician, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study.
* Have shown a previous immediate hypersensitivity response, including anaphylaxis, to an immunoglobulin product (plasma-derived or recombinant, e.g., monoclonal antibody).
* Have a known allergy to murine proteins or other chimeric proteins.
* Have or have had any of the following infections within 6 months of screening: herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB.
* Have a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to screening).
* Have a concomitant diagnosis or any history of congestive heart failure (CHF).
* History of noncompliance to medical regimens, or other condition/circumstance that could interfere with the patient's adherence to protocol requirements (e.g., psychiatric disease, lack of motivation, travel, etc).
* Any cause of liver disease other than chronic hepatitis C, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Non-alcoholic steatohepatitis (NASH)
  * Drug-related liver disease
* Subject with a positive TST might be enrolled if the diagnosis of tuberculosis is ruled out. To rule out TB, the following criteria must be met:
* The medical history is negative for symptoms of TB
* The physical examination must reveal no observations that could be related to TB
* The patient has a documented adequate course of treatment for either LTBI or TB at least 6 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-07-18 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have achieved sustained virological response (SVR) in the infliximab (induction dose) plus PEGETRON and the PEGETRON groups at 24 weeks post treatment end | 24 weeks after completion of up to 48 weeks of PEGETRON therapy

SECONDARY OUTCOMES:
Early virological response (EVR) | Week 12 of PEGETRON treatment period
Safety parameters | During 48-week PEGETRON treatment period and 24-week follow up

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php